CLINICAL TRIAL: NCT04726579
Title: An Open-Label, Prospective, Observational Study to Assess the Response to Cannabidiol (CBD) Oil in Subjects With Chronic Mechanical Back Pain (MBP)
Brief Title: CBD Oil in Mechanical Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: perceiveMD (Other)
Responsible Party: Principal Investigator, Jonathan Chan, Principal Investigator, perceiveMD
Other Study IDs: H20-02124
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a 12-week open-label, prospective, observational study to assess how subjects with chronic mechanical back pain respond to cannabidiol (CBD)

DETAILED DESCRIPTION:
Purpose: To Assess the Response to Cannabidiol (CBD) Oil in Subjects with Chronic Mechanical Back Pain (MBP)

Hypothesis: Cannabis use provides many patients with significant low back pain relief.

Justification: Mechanical back pain is a condition affecting around 30% of the general adult population. It is the second most common reason to see a family physician and the most common reason patients end up on work disability. Long term chronic pain is associated with mood and anxiety disorders in a lot of patients, which suggests that a successful plan for the treatment of chronic pain must also consider the treatment of possible co-existing psychiatrist conditions.

Objectives:

To assess the change in pain measured by 0 to 10 point visual analogue scale (VAS) for patients with chronic mechanical back pain treated with CBD oil

Research Design:

52 patients with pain severity ≥4/10 on Visual Analog Scale (VAS) for at least 3 months who have decided to take CBD oil (up to 50 mg SL BID) to manage their symptoms will be recruited to participate. As per standard of care, patients will be encouraged to keep baseline doses of analgesics (if any) stable for the first 6 weeks of the study to monitor their response to CBD oil. Analgesic medications will be allowed to be adjusted between weeks 6 to 12.

Enrolled patients will be assessed at baseline, week 6, and week 12 for a total of 3 virtual visits. Patients will be asked to fill out online questionnaires and a medication diary to assess effectiveness and compliance. Safety will also be assessed throughout the study. Patients will be asked to report any adverse events (AEs) at study completion or earlier if they decide to withdraw. In addition, they will be provided a phone number to PerceiveMD where they can report any serious adverse events (SAEs) in between scheduled visits. Patients will be instructed to report any SAEs within 24 hours. PerceiveMD will then communicate this to one of the Investigators the same day. All adverse reactions will be recorded in the study electronic medical record (EMR), InputHealth.

Statistical Analysis:

The primary analysis will be measured in all enrolled patients who are dispensed drug. Patient data will be collected using online electronic questionnaires generated through InputHealth and stored within InputHealth. Patient data will additionally be collected at the time of their virtual visits with the Investigator(s) at PerceiveMD. This data will be recorded and stored within InputHealth. For descriptive summaries, the mean, sample size (n), standard deviation (SD), standard error (SE), median, minimum (min), and maximum (max) will be calculated for continuous variables. For categorical variables, frequency and percentage in each category will be provided. Change from baseline value will be calculated at each visit. No imputation will be made for missing values. Pain VAS, modified Oswestry Low Back Pain Disability, and GAD7 will be compared between groups, with mean values and 95% confidence interval provided. Percentage of patients with 30% and 50% improvement in pain VAS will also be assessed. Change in analgesic medication dose and use will be analyzed and reported. Based on the extent of missing data, additional analyses may be conducted (e.g. last observation carried forward (LOCF), non-responder index) as a sensitivity analysis to support the primary analysis

ELIGIBILITY:
Inclusion Criteria:

1) Must be able to communicate well with the Investigator(s), understand and comply with the requirements of the study, and provide written consent

2. Age ≥21 years

3. Diagnosed with MBP with symptom onset >3 months prior to screening visit

4. Must have pain severity ≥4/10 on VAS for at least 3 months as reported by the patient

5. Decided to take CBD oil for the treatment of MBP

6. Must have access to a computer or laptop and be able to operate the required video conference platform

Exclusion Criteria:

* 1. Cause of pain due to malignancy, infection, fracture, or spondylarthritis

  2. Recent (within the last 3 months) spinal trauma

  3. Leg dominant/radicular pain

  4. Current active fibromyalgia

  5. Female who is pregnant, nursing, or plan to become pregnant during the study

  6. Allergies to CBD or any components of the CBD oil to be used in the study

  7. Active significant medical and/or psychological illness which, in the opinion of the Investigator,

is not suitable to participate in the study (e.g. malignancy, hepatic disease, CAD, COPD, schizophrenia, etc.)

8. Changes in doses of baseline analgesics such as acetaminophen, pregabalin, gabapentin, opioids, or glucocorticoids within 1 month prior to the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. This study will be based out of PerceiveMD, a clinic with expertise in CBD therapy. Patients will be approached for enrollment at rheumatology, physiatry, and pain clinics as well as PerceiveMD.
     Baseline screening visit and follow will be done online using a PIPA/PIPEDA compliant video or audio conference. Prospective patients are those who have decided to take CBD oil for the treatment of MBP.
  2. Flyers will be given to health care providers at rheumatology, physiatry, and pain clinics as well as PerceiveMD. Flyers will also be directly available to patients at these locations and they can contact Dr. Lim if they would like to participate in the study.
  3. Prospective patients will be identified using the following criteria:
     Equal to or older than 21 years old Back pain for more than 3 months (self-reported) prior to screening visit
  4. The study will be conducted at PerceiveMD, 603 Gorge Rd. E Victoria, BC
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the change in pain measured by 0 to 10 point visual analogue scale (VAS) for patients with chronic mechanical back pain treated with CBD oil | 12 weeks
  52 patients with pain severity ≥4/10 on Visual Analog Scale (VAS) for at least 3 months who have decided to take CBD oil (up to 50 mg SL BID) to manage their symptoms will be recruited to participate. As per standard of care, patients will be encouraged to keep baseline doses of analgesics (if any) stable for the first 6 weeks of the study to monitor their response to CBD oil. Analgesic medications will be allowed to be adjusted between weeks 6 to 12.